CLINICAL TRIAL: NCT01243671
Title: A Multi-Center Study of Adalimumab in Japanese Subjects With Intestinal Behçet's Disease
Brief Title: A Study of Adalimumab in Japanese Subjects With Intestinal Behçet's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M11-509
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Results first posted 2013-05-15 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-06

CONDITIONS: Intestinal Behçet's Disease
Keywords: Behçet's, intestinal
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab (Experimental): Adalimumab 160 mg at Week 0, 80 mg at Week 2 and 40 mg every other week (eow) starting at Week 4 to Week 50, subcutaneous injection. After Week 52, participants could continue the treatment with 40 mg eow until the day before approval of adalimumab for intestinal Behçet's disease in Japan.
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab
  Other Names: ABT-D2E7, Humira

SUMMARY:
To investigate efficacy, safety and pharmacokinetics of adalimumab subcutaneous (sc) for Japanese subjects with intestinal Behçet's disease who are refractory to conventional therapies.

ELIGIBILITY:
Inclusion Criteria:

* Intestinal Behçet's disease
* Patients with typical ulcer at ileocecal region
* Patients who have failed conventional treatment

Exclusion Criteria:

* Crohn's disease
* History of ileocecal resection
* History of tuberculosis (TB)
* Female subject who is pregnant or breast-feeding or considering becoming pregnant during the study

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morio Ozawa, MS, Study Director — AbbVie
Locations (12):
- Japan (12):
  - Site Reference ID/Investigator# 46738, Chikushino-shi
  - Site Reference ID/Investigator# 46723, Kurume
  - Site Reference ID/Investigator# 46728, Nagoya
  - Site Reference ID/Investigator# 46725, Nishinomiya-shi
  - Site Reference ID/Investigator# 46730, Osaka
  - Site Reference ID/Investigator# 46722, Sagamihara-shi
  - Site Reference ID/Investigator# 46726, Sakura
  - Site Reference ID/Investigator# 59578, Sapporo
  - Site Reference ID/Investigator# 46724, Takatsuki-shi
  - Site Reference ID/Investigator# 46729, Tokyo
  - Site Reference ID/Investigator# 46737, Tokyo
  - Site Reference ID/Investigator# 46733, Yokohama

REFERENCES:
- [Derived] Inoue N, Kobayashi K, Naganuma M, Hirai F, Ozawa M, Arikan D, Huang B, Robinson AM, Thakkar RB, Hibi T. Long-term safety and efficacy of adalimumab for intestinal Behcet's disease in the open label study following a phase 3 clinical trial. Intest Res. 2017 Jul;15(3):395-401. doi: 10.5217/ir.2017.15.3.395. Epub 2017 Jun 12. PMID 28670237
- [Derived] Tanida S, Inoue N, Kobayashi K, Naganuma M, Hirai F, Iizuka B, Watanabe K, Mitsuyama K, Inoue T, Ishigatsubo Y, Suzuki Y, Nagahori M, Motoya S, Nakamura S, Arora V, Robinson AM, Thakkar RB, Hibi T. Adalimumab for the treatment of Japanese patients with intestinal Behcet's disease. Clin Gastroenterol Hepatol. 2015 May;13(5):940-8.e3. doi: 10.1016/j.cgh.2014.08.042. Epub 2014 Sep 19. PMID 25245624
- See also: Related info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adalimumab
Started | 20
Completed 24 Weeks of Treatment | 18
Completed 52 Weeks of Treatment | 17
Completed | 15 (Completed 136 weeks of treatment.)
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Anti-adalimumab antibody positive | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (13.33)
Age, Customized [Number; unit: participants]
  <40 years | 11
  Between 40 and 65 years | 7
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Longest Diameter of Ileocecal Largest Open Ulcer [Number; unit: participants] — Number of participants with longest diameter of ileocecal largest open ulcer in each of 3 categories, as determined by screening (baseline) endoscopy.
  participants
    >=1 cm to <2 cm | 8
    >=2 cm to <3 cm | 5
    >=3 cm | 7
Global Assessment of Gastrointestinal (GI) Symptoms Grade [Number; unit: participants] — Global assessment of gastrointestinal symptoms is a participant-assessed, investigator-confirmed grading of global symptoms from 0 to 4: 0=free of symptoms; 1=symptoms existed in past 2 weeks but did not affect participant's daily life; 2=symptoms existed in past 2 weeks and slightly affected participant's daily life; 3=symptoms existed in past 2 weeks and affected participant's daily life; 4=symptoms existed in past 2 weeks and critically affected participant's daily life.
  participants
    Grade 0 | 0
    Grade 1 | 0
    Grade 2 | 0
    Grade 3 | 15
    Grade 4 | 5
Assessment of Abdominal Pain (GI Symptom Component) Grade [Number; unit: participants] — Assessment of gastrointestinal symptom component of abdominal pain via a participant-assessed, investigator-confirmed grading of symptoms from 0 to 4: 0=free of symptoms; 1=symptoms existed in past 2 weeks but did not affect participant's daily life; 2=symptoms existed in past 2 weeks and slightly affected participant's daily life; 3=symptoms existed in past 2 weeks and affected participant's daily life; 4=symptoms existed in past 2 weeks and critically affected participant's daily life.
  participants
    Grade 0 | 2
    Grade 1 | 1
    Grade 2 | 3
    Grade 3 | 10
    Grade 4 | 4
Assessment of Diarrhea (GI Symptom Component) Grade [Number; unit: participants] — Assessment of gastrointestinal symptom component of diarrhea via a participant-assessed, investigator-confirmed grading of symptoms from 0 to 4: 0=free of symptoms; 1=symptoms existed in past 2 weeks but did not affect participant's daily life; 2=symptoms existed in past 2 weeks and slightly affected participant's daily life; 3=symptoms existed in past 2 weeks and affected participant's daily life; 4=symptoms existed in past 2 weeks and critically affected participant's daily life.
  participants
    Grade 0 | 4
    Grade 1 | 6
    Grade 2 | 0
    Grade 3 | 9
    Grade 4 | 1
Assessment of Other Symptoms (GI Symptom Component) Grade [Number; unit: participants] — Assessment of gastrointestinal symptoms other than abdominal pain or diarrhea (abdominal discomfort/fullness, etc) via a participant-assessed, investigator-confirmed grading of symptoms from 0 to 4: 0=free of symptoms; 1=symptoms existed in past 2 weeks but did not affect participant's daily life; 2=symptoms existed in past 2 weeks and slightly affected participant's daily life; 3=symptoms existed in past 2 weeks and affected participant's daily life; 4=symptoms existed in past 2 weeks and critically affected participant's daily life. Scores assess symptoms in the 2 weeks prior to Baseline.
  participants
    Grade 0 | 0
    Grade 1 | 1
    Grade 2 | 4
    Grade 3 | 12
    Grade 4 | 3
Assessment of Behçet's Disease Symptoms (Other Than GI Symptoms) Grade [Number; unit: participants] — Investigators assessed oral aphthous, skin symptoms (erythema nodosum rash), eye symptoms (uveitis) and vulval (genital) ulcers during 4 weeks before baseline visit via participant interview at baseline, using the following grades: 0=None; 1=Symptom existed less than 2 weeks, or 1 eye crisis in recent 4 weeks; 2=Symptom existed 2 weeks or more, or 2 eye crises in recent 4 weeks; 3=Symptom existed mostly in recent 4 weeks, or 3 eye crises in recent 4 weeks.
  participants
    Oral Aphthous Grade 0 | 5
    Oral Aphthous Grade 1 | 8
    Oral Aphthous Grade 2 | 3
    Oral Aphthous Grade 3 | 4
    Skin (Erythema Nodosum Rash) Grade 0 | 12
    Skin (Erythema Nodosum Rash) Grade 1 | 4
    Skin (Erythema Nodosum Rash) Grade 2 | 1
    Skin (Erythema Nodosum Rash) Grade 3 | 3
    Eye (Uveitis) Grade 0 | 20
    Eye (Uveitis) Grade 1 | 0
    Eye (Uveitis) Grade 2 | 0
    Eye (Uveitis) Grade 3 | 0
    Vulval (Genital) Ulcer Grade 0 | 17
    Vulval (Genital) Ulcer Grade 1 | 1
    Vulval (Genital) Ulcer Grade 2 | 0
    Vulval (Genital) Ulcer Grade 3 | 2
Inflammatory Bowel Disease Questionnaire (IBDQ) [Mean (Standard Deviation); unit: units on a scale] — Inflammatory Bowel Disease Questionnaire (IBDQ) is the standard questionnaire to assess the quality of life of patients with inflammatory bowel disease. The IBDQ is a 32-item questionnaire consisting of 4 dimensions: bowel-related symptoms, systemic function, social function, and emotional status. The responses to each question within each domain range from 1 (significant impairment) to 7 (no impairment), with total score ranging from 32 (very poor) to 224 (perfect health-related quality of life).
  units on a scale | 140.5 (36.18)
Short-Form-36 (SF-36) Summary Scores [Mean (Standard Deviation); unit: units on a scale] — The Short-Form-36 (SF-36) Health Survey is a comprehensive quality of life scale. An increase in SF-36 score indicates alleviation of the disease and a decrease in score indicates aggravation of disease. The physical component reflects activity level, activity limitations, pain, and rating of one's health. Score on the physical component ranges from 0 (poorest health) to 100 (best health). The mental component reflects vitality, social functioning, role-emotional, and mental health. Score on the mental component ranges from 0 (poorest health) to 100 (best health).
  units on a scale
    Physical Component Summary | 41.8 (5.70)
    Mental Component Summary | 34.6 (12.43)
C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: mg/dL] — C-Reactive Protein (CRP) normal range was defined as ≤0.3 mg/dL.
  mg/dL | 0.8 (1.17)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Marked Improvement at Week 24
Description: Marked improvement is defined as the combination of both global assessment of gastrointestinal (GI) symptoms and endoscopic improvement grades of ≤1. Global assessment of GI symptoms is a participant-assessed, investigator-confirmed grading of global symptoms from 0 to 4: 0=free of symptoms; 1=symptoms existed in past 2 weeks but did not affect participant's daily life; 2=symptoms existed in past 2 weeks and slightly affected participant's daily life; 3=symptoms existed in past 2 weeks and affected participant's daily life; 4=symptoms existed in past 2 weeks and critically affected participant's daily life. Endoscopic improvement was assessed in 4 grades compared to the screening endoscopy based on the longest diameter (none, ≥1 cm to <2 cm, ≥2 cm to <3 cm, ≥3 cm) of ileocecal largest open ulcer (area of mucosal defect). Grades are: 0=healing; 1=marked reduction (reduction to ≤1/4); 2=reduction (reduction to ≤1/2 - 1/4); 3=no change or worse (reduction less than 1/2 or expansion).
Time Frame: 24 weeks
Population: Full analysis set (all participants). Those with missing evaluations were imputed as non-responders.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 20
participants | 9

2. Secondary Outcome: Number of Participants With Marked Improvement at Week 52
Description: as for outcome 1
Time Frame: 52 weeks
Population: Full analysis set (all participants). Those with missing evaluations were imputed as non-responders.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 20
participants | 12

3. Secondary Outcome: Number of Participants With Complete Remission at Week 24 and Week 52
Description: Complete remission was defined as both endoscopic improvement and global assessment of gastrointestinal symptoms grades of 0. Endoscopic improvement was assessed in 4 grades compared to the screening (baseline) endoscopy based on the longest diameter (none, ≥1 cm to <2 cm, ≥2 cm to <3 cm, ≥3 cm) of ileocecal largest open ulcer (area of mucosal defect). Grades are: 0=healing; 1=marked reduction (reduction to ≤1/4); 2=reduction (reduction to ≤1/2 - 1/4); 3=no change or worse (reduction less than 1/2 or expansion). Global assessment of gastrointestinal symptoms is a participant-assessed, investigator-confirmed grading of global symptoms from 0 to 4: 0=free of symptoms; 1=symptoms existed in past 2 weeks but did not affect participant's daily life; 2=symptoms existed in past 2 weeks and slightly affected participant's daily life; 3=symptoms existed in past 2 weeks and affected participant's daily life; 4=symptoms existed in past 2 weeks and critically affected participant's daily life.
Time Frame: 24 weeks, 52 weeks
Population: Full analysis set (all participants). Those with missing evaluations were imputed as non-responders.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 20
participants
  Week 24 | 4
  Week 52 | 4

4. Secondary Outcome: Number of Participants With a Global Assessment of Gastrointestinal Symptoms Grade 0 or ≤1 and Improvement of ≥1 Grade at Week 24 and Week 52
Description: Study participants completed a global assessment of their gastrointestinal symptoms (Behçet's disease symptoms other than gastrointestinal symptoms were excluded) during 2 weeks before assessment visit on a 5-grade scale. The investigator confirmed this assessment via interview with participants. Assessment is graded from 0 to 4: 0=free of symptoms; 1=symptoms existed in past 2 weeks but did not affect participant's daily life; 2=symptoms existed in past 2 weeks and slightly affected participant's daily life; 3=symptoms existed in past 2 weeks and affected participant's daily life; 4=symptoms existed in past 2 weeks and critically affected participant's daily life. Global assessment of grade 0 or ≤1 and improvement of ≥1 (from baseline) is presented.
Time Frame: 24 weeks, 52 weeks
Population: Full analysis set (all participants). Those with missing evaluations were imputed as non-responders.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 20
participants
  Week 24: Grade 0 | 9
  Week 24: Grade ≤1 | 13
  Week 24: Improvement of ≥1 Grade | 16
  Week 52: Grade 0 | 9
  Week 52: Grade ≤1 | 16
  Week 52: Improvement of ≥1 Grade | 18

5. Secondary Outcome: Number of Participants With Endoscopic Improvement Grades 0, ≤1 and ≤2 at Week 24 and Week 52
Description: Endoscopic improvement was assessed in 4 grades compared to the screening (baseline) endoscopy based on the longest diameter (none, ≥1 cm to <2 cm, ≥2 cm to <3 cm, ≥3 cm) of ileocecal largest open ulcer (area of mucosal defect). Grades are: 0=healing; 1=marked reduction (reduction to ≤1/4); 2=reduction (reduction to ≤1/2 - 1/4); 3=no change or worse (reduction less than 1/2 or expansion).
Time Frame: 24 weeks, 52 weeks
Population: Full analysis set (all participants). Those with missing evaluations were imputed as non-responders.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 20
participants
  Week 24: Grade 0 | 9
  Week 24: Grade ≤1 | 12
  Week 24: Grade ≤2 | 15
  Week 52: Grade 0 | 11
  Week 52: Grade ≤1 | 13
  Week 52: Grade ≤2 | 15

6. Secondary Outcome: Number of Participants With Abdominal Pain, Diarrhea and Other Gastrointestinal (GI) Symptoms Grade ≤1 and Improvement of ≥1 Grade at Week 24 and Week 52
Description: Participants assessed their abdominal pain, diarrhea and other gastrointestinal symptoms (abdominal discomfort, abdominal fullness, etc) during 2 weeks before assessment visit in 5 grades. Investigator confirmed the assessment through interview with participants. Assessment is graded from 0 to 4: 0=free of symptoms; 1=symptoms existed in past 2 weeks but did not affect participant's daily life; 2=symptoms existed in past 2 weeks and slightly affected participant's daily life; 3=symptoms existed in past 2 weeks and affected participant's daily life; 4=symptoms existed in past 2 weeks and critically affected participant's daily life. Improvement of ≥1 grade from baseline is also presented.
Time Frame: 24 weeks, 52 weeks
Population: Full analysis set (all participants). n=number of participants who had any symptom at baseline. Those with missing evaluations were imputed as non-responders.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 20
participants
  Week 24: Abdominal Pain Grade ≤1; n=18 | 11
  Week 24: Diarrhea Grade ≤1; n=16 | 13
  Week 24: Other GI Symptom Grade ≤1; n=20 | 16
  Week 24:Abdominal Pain Improvement ≥1 Grade; n=18 | 14
  Week 24: Diarrhea Improvement ≥1 Grade; n=16 | 11
  Week 24:Other GI Symptom Improvement ≥1 Grade;n=20 | 18
  Week 52: Abdominal Pain Grade ≤1; n=18 | 14
  Week 52: Diarrhea Grade ≤1; n=16 | 15
  Week 52: Other GI Symptom Grade ≤1; n=20 | 16
  Week 52:Abdominal Pain Improvement ≥1 Grade; n=18 | 16
  Week 52: Diarrhea Improvement ≥1 Grade; n=16 | 13
  Week 52:Other GI Symptom Improvement ≥1 Grade;n=20 | 18

7. Secondary Outcome: Number of Participants With Resolution of Behçet's Disease Symptoms (Other Than Gastrointestinal Symptoms) at Week 24 and Week 52
Description: Investigators assessed oral aphthous (mouth ulcers), skin symptoms, eye symptoms and vulval (genital) ulcers during 4 weeks before study visit via participant interview, using the following grades. Oral aphthous: 0=None; 1=Symptom existed less than 2 weeks in recent 4 weeks; 2=Symptom existed 2 weeks or more in recent 4 weeks; 3=Symptom existed mostly in recent 4 weeks. Skin (Erythema nodosum rash): 0=None; 1=Symptom existed less than 2 weeks in recent 4 weeks; 2=Symptom existed 2 weeks or more in recent 4 weeks; 3=Symptom existed mostly in recent 4 weeks. Eye (Uveitis): 0=None; 1=one eye crisis in recent 4 weeks; 2=two eye crises in recent 4 weeks; 3=three eye crises in recent 4 weeks. Vulval (genital) ulcer: 0=None; 1=Symptom existed less than 2 weeks in recent 4 weeks; 2=Symptom existed 2 weeks or more in recent 4 weeks; 3=Symptom existed mostly in recent 4 weeks. Resolution was defined as: Behçet's disease symptoms other than gastrointestinal symptoms were graded 0 (disappeared).
Time Frame: 24 weeks, 52 weeks
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 20
participants
  Week 24: Oral Aphthous; n=15 | 10
  Week 24: Skin (Erythema nodosum rash); n=8 | 6
  Week 24: Eye (Uveitis); n=0 | 0
  Week 24: Vulval (Genital) Ulcer; n=3 | 2
  Week 52: Oral Aphthous; n=15 | 10
  Week 52: Skin (Erythema nodosum rash); n=8 | 7
  Week 52: Eye (Uveitis); n=0 | 0
  Week 52: Vulval (Genital) Ulcer; n=3 | 2

8. Secondary Outcome: Mean Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) at Week 24 and Week 52
Description: Inflammatory Bowel Disease Questionnaire (IBDQ) is the standard questionnaire to assess the quality of life of patients with inflammatory bowel disease. The IBDQ is a 32-item questionnaire consisting of 4 dimensions: bowel-related symptoms, systemic function, social function and emotional status. The responses to each question within each domain range from 1 (significant impairment) to 7 (no impairment), with total score ranging from 32 (very poor) to 224 (perfect health-related quality of life).
Time Frame: Baseline, 24 weeks, 52 weeks
Population: Full analysis set (all participants). Those with missing evaluations were imputed by last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 20
units on a scale
  Week 24 | 37.1 (40.00)
  Week 52 | 41.2 (41.91)

9. Secondary Outcome: Mean Change From Baseline in Short Form-36 (SF-36) Summary Scores at Week 24 and Week 52
Description: The Short-Form-36 (SF-36) Health Survey is a comprehensive quality of life scale. An increase in SF-36 score indicates alleviation of the disease and a decrease in score indicates aggravation of disease. The physical component reflects activity level, activity limitations, pain and rating of one's health. Score on the physical component ranges from 0 (poorest health) to 100 (best health). The mental component reflects vitality, social functioning, role-emotional and mental health. Score on the mental component ranges from 0 (poorest health) to 100 (best health).
Time Frame: Baseline, 24 weeks, 52 weeks
Population: Full analysis set (all participants). Those with missing evaluations were imputed by last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 20
units on a scale
  Week 24: Summary Score (Physical Component) | 7.5 (7.18)
  Week 24: Summary Score (Mental Component) | 8.9 (12.85)
  Week 52: Summary Score (Physical Component) | 9.0 (8.42)
  Week 52: Summary Score (Mental Component) | 9.0 (13.27)

10. Secondary Outcome: Median Change From Baseline in C-Reactive Protein (CRP) at Week 24 and Week 52
Description: C-Reactive Protein (CRP) normal range was defined as ≤0.3 mg/dL.
Time Frame: Baseline, 24 weeks, 52 weeks
Population: Full analysis set (all participants). Those with missing evaluations were imputed by last observation carried forward.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Adalimumab
Number analyzed (Participants) | 20
mg/dL
  Week 24 | -0.3 (1.27) [-3.0 to 3.0]
  Week 52 | -0.2 (2.22)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were reported from the time of study drug administration up to 124 weeks + 70 days following discontinuation of study drug. Serious AEs were collected from the time the participant signed the study-specific informed consent.
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 6/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=20)
AUTOIMMUNE THYROIDITIS (Endocrine disorders) | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
SUBILEUS (Gastrointestinal disorders) | 1
BEHCET'S SYNDROME (Immune system disorders) | 1
ABSCESS INTESTINAL (Infections and infestations) | 1
APPENDICITIS (Infections and infestations) | 1
APPENDICITIS PERFORATED (Infections and infestations) | 1
SPONDYLITIC MYELOPATHY (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=20)
ANAEMIA (Blood and lymphatic system disorders) | 1
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1
SYRINGOMYELIA (Congenital, familial and genetic disorders) | 1
BLEPHARITIS (Eye disorders) | 1
CHALAZION (Eye disorders) | 1
CONJUNCTIVITIS (Eye disorders) | 1
DRY EYE (Eye disorders) | 1
OCULAR HYPERAEMIA (Eye disorders) | 1
VISION BLURRED (Eye disorders) | 1
VITREOUS FLOATERS (Eye disorders) | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
CHEILITIS (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
DENTAL CARIES (Gastrointestinal disorders) | 3
DIARRHOEA (Gastrointestinal disorders) | 3
ENTEROCOLITIS (Gastrointestinal disorders) | 1
GASTRIC POLYPS (Gastrointestinal disorders) | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 2
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 1
ORAL DISORDER (Gastrointestinal disorders) | 1
PALATAL OEDEMA (Gastrointestinal disorders) | 1
PROCTITIS (Gastrointestinal disorders) | 1
SMALL INTESTINE ULCER (Gastrointestinal disorders) | 1
STOMATITIS (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
FOREIGN BODY REACTION (General disorders) | 1
GRANULOMA (General disorders) | 1
INJECTION SITE REACTION (General disorders) | 2
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1
LIVER DISORDER (Hepatobiliary disorders) | 1
BEHCET'S SYNDROME (Immune system disorders) | 3
ACUTE TONSILLITIS (Infections and infestations) | 1
BACTERIAL INFECTION (Infections and infestations) | 1
BRONCHITIS (Infections and infestations) | 1
CAMPYLOBACTER INFECTION (Infections and infestations) | 1
CYSTITIS (Infections and infestations) | 1
ENTERITIS INFECTIOUS (Infections and infestations) | 2
FURUNCLE (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 3
GASTROENTERITIS VIRAL (Infections and infestations) | 1
GINGIVITIS (Infections and infestations) | 1
HERPES ZOSTER (Infections and infestations) | 1
HORDEOLUM (Infections and infestations) | 2
INFLUENZA (Infections and infestations) | 2
NASOPHARYNGITIS (Infections and infestations) | 11
ORAL HERPES (Infections and infestations) | 2
OTITIS MEDIA (Infections and infestations) | 1
PHARYNGITIS (Infections and infestations) | 2
TINEA INFECTION (Infections and infestations) | 1
TINEA VERSICOLOUR (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
ARTHROPOD STING (Injury, poisoning and procedural complications) | 1
CONTUSION (Injury, poisoning and procedural complications) | 3
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1
ANTINUCLEAR ANTIBODY INCREASED (Investigations) | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1
BLOOD CHOLESTEROL INCREASED (Investigations) | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1
CARCINOEMBRYONIC ANTIGEN INCREASED (Investigations) | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1
MYCOBACTERIUM TUBERCULOSIS COMPLEX TEST POSITIVE (Investigations) | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1
OBESITY (Metabolism and nutrition disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2
BENIGN NEOPLASM OF THYROID GLAND (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
RECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
DIZZINESS (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 5
HYPOAESTHESIA (Nervous system disorders) | 1
LACUNAR INFARCTION (Nervous system disorders) | 1
AFFECTIVE DISORDER (Psychiatric disorders) | 1
INSOMNIA (Psychiatric disorders) | 1
HYPERTONIC BLADDER (Renal and urinary disorders) | 1
DYSMENORRHOEA (Reproductive system and breast disorders) | 1
PROSTATIC CYST (Reproductive system and breast disorders) | 1
UTERINE POLYP (Reproductive system and breast disorders) | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 4
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1
ACNE (Skin and subcutaneous tissue disorders) | 2
DERMATITIS (Skin and subcutaneous tissue disorders) | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 2
ECZEMA NUMMULAR (Skin and subcutaneous tissue disorders) | 1
PAPULE (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 3
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1
SKIN MASS (Skin and subcutaneous tissue disorders) | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 2
HYPERTENSION (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.